CLINICAL TRIAL: NCT00326469
Title: Phase II, Open, Single Group, Multicentre Study to Evaluate the Efficacy and Safety of Lanreotide Autogel Administered Every 4 Weeks by Deep Subcutaneous Injection in the Tumour's Growth Stabilization of Patients With Progressive Neuroendocrine Tumours Who Are Not Eligible to be Treated With Either Surgery or Chemotherapy
Brief Title: Efficacy and Safety of Lanreotide Autogel in Tumour Stabilization of Patients With Progressive Neuroendocrine Tumours
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A-92-52030-166; 2004-002871-18 (EudraCT Number)
Record Dates: First submitted 2006-05-15; First posted 2006-05-16 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Neuroendocrine Tumours
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — lanreotide

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: lanreotide (Autogel formulation)

INTERVENTIONS:
Drug: lanreotide (Autogel formulation) — 120mg administered via deep subcutaneous injection every 28 days for up to 24 months or until disease progression.

SUMMARY:
To evaluate, in patients with progressive neuroendocrine tumours who are not eligible to be treated with either surgery or chemotherapy at the moment of study inclusion, the efficacy of lanreotide Autogel in tumour growth stabilization.

ELIGIBILITY:
Inclusion Criteria:

* patients with histopathologic diagnosis of well-differentiated neuroendocrine tumour or carcinoma according to WHO classification
* patients who, according to RECIST criteria (Response Evaluation Criteria in Solid Tumours) present measurable disease
* patients with progressive disease in the previous 6 months before their inclusion in the study
* patients with positive IN111 octreotide scintigraphy

Exclusion Criteria:

* patients with surgically removable localised disease
* patients with progressive disease in the first six months of being diagnosed
* patients with intestinal obstruction due to a carcinoid tumour
* patients who have received treatment with somatostatin analogues during the 6 months before being included in the study
* patients who have received treatment with radiotherapy, chemotherapy or interferon 4 weeks before being included in the study, or planned to receive these during the study
* patients who have received treatment with liver artery embolisation or radiopharmaceuticals (endoradiotherapy) 12 weeks before being included in the study, or planned during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-05; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Time to disease progression (appearance of 1+ new lesions or increase >or= to 20% of sum of the longest diameters of target lesions compared to the lower sum of maximum diameters recorded since the start of the study). | Month 3, 6, 9, 12, 15, 18, 21 and 24

SECONDARY OUTCOMES:
To evaluate efficacy related to tumour's partial or total response, biological disease markers response, symptomatic control, effect of treatment on patient's quality of life | Month 3, 6, 9, 12, 15, 18, 21 and 24
Identify tumour growth stabilization predictive factors under treatment with lanreotide Autogel | Month 3, 6, 9, 12, 18, 21 and 24
Tolerance | All visits

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (27):
- Spain (27):
  - H. Juan Canalejo, A Coruña
  - H. Virgen de los Lirios, Alcoy
  - H. General Univ. de Alicante, Alicante
  - H. Germans Trias i Pujol, Badalona
  - H. Santa Creu i Sant Pau, Barcelona
  - H. Clínic i Provincial, Barcelona
  - Corporación H. Parc Tauli, Barcelona
  - Consorci Sanitari de Terrassa, Barcelona
  - H. General de Hospitalet, Barcelona
  - H. de Basurto, Bilbao
  - H. General de Elche, Elche
  - H. de la Princesa, Madrid
  - H. Ramón y Cajal, Madrid
  - H. Clínico Univ. San Carlos, Madrid
  - H. 12 de Octubre, Madrid
  - H. Severo Ochoa, Madrid
  - Fundación H. Son Llàtzer, Palma de Mallorca
  - Consorcio H. de Pontevedre, Pontevedra
  - H. de Sagunto, Sagunto
  - H. Clínico de Salamanca, Salamanca
  - Int. Oncológico San Sebastián, San Sebastián
  - H. Univ. de Canarias, Santa Cruz de Tenerife
  - H. Marques de Valdecilla, Santander
  - Hospital Universitario "Dr. Peset", Valencia
  - H. La Fe, Valencia
  - H. Hospital General Universitario de Valencia, Valencia
  - H. Miguel Servet, Zaragoza

REFERENCES:
- [Derived] Martin-Richard M, Massuti B, Pineda E, Alonso V, Marmol M, Castellano D, Fonseca E, Galan A, Llanos M, Sala MA, Pericay C, Rivera F, Sastre J, Segura A, Quindos M, Maisonobe P; TTD (Tumores del Tracto Digestivo) Study Group. Antiproliferative effects of lanreotide autogel in patients with progressive, well-differentiated neuroendocrine tumours: a Spanish, multicentre, open-label, single arm phase II study. BMC Cancer. 2013 Sep 20;13:427. doi: 10.1186/1471-2407-13-427. PMID 24053191